CLINICAL TRIAL: NCT04233736
Title: Bilateral Erector Spinae Plane Blocks (ESP) for Postoperative Pain in Lumbo-sacral Spine Surgery: A Double-blinded Randomized Controlled Trial
Brief Title: Erector Spinae Plane Blocks (ESP) for Postoperative Pain in Lumbo-sacral Spine Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-28625
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Erector Spinae Plane Block; Lumbar Spine Surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Active Comparator)
  Interventions: Procedure: Bilateral lumbar erector spinae plane block
- Control group (Sham Comparator)
  Interventions: Procedure: Bilateral lumbar erector spinae plane block

INTERVENTIONS:
Procedure: Bilateral lumbar erector spinae plane block — Bilateral lumbar erector spinae plane blocks performed under ultrasound guidance

SUMMARY:
The goal of this study is to evaluate the analgesic efficacy of bilateral erector spinae plane (ESP) blocks after lumbar and lumbo-sacral spine surgery by assessing postoperative pain scores and opiate requirements as the primary outcome measures. We are aiming to investigate how ESP blocks, performed under ultrasound guidance at the T12 vertebral level, contribute to postoperative pain control. This will be determined by measuring numerical rating pain scores repeatedly following surgery and opiate consumption until patient discharge from hospital. These primary outcome measures will be compared between a treatment group of participants, who will receive ESP blocks and a control group who will receive a sham block. Our primary hypothesis is that ESP blocks significantly reduce postoperative pain and opiate requirements

ELIGIBILITY:
Inclusion Criteria:

* Spine surgery at or below the L1 vertebral level
* Midline surgical approach

Exclusion Criteria:

* Previous lumbar or lumbo-sacral surgery with or without hardware placement
* Evidence of dura pathology (including CSF leak)
* Spine tumor
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain scores | During hospitalization, typically lasting between 1 and 5 days
  Pain scores will be measured and documented as part of routine clinical care using the standard NRS (numerical rating scale, ranging from 0= no pain to 10= worst imaginable pain). Pain assessments will be made several times per day starting pre-operatively and continued during hospitalization.
Perioperative opiate consumption | During hospitalization, typically lasting between 1 and 5 days
  Peri-operative opiate consumption will be assessed by measuring opiate administration intra- and post-operatively (during hospitalization) and expressed as oral morphine equivalents (OMEs).

CONTACTS AND LOCATIONS:
Overall Officials: Claas Siegmueller, MD PhD MBA, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No